CLINICAL TRIAL: NCT04587479
Title: A Phase 1, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-8263 in Adult Subjects With Advanced Solid Tumors
Brief Title: A First-in-Human Study of JAB-8263 in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAB-8263-1001
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors, Adult
Keywords: BET inhibitor; Bromodomain and Extra-terminal

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JAB-8263 (Experimental): Monotherapy, dose escalation
  Interventions: Drug: JAB-8263

INTERVENTIONS:
Drug: JAB-8263 — Variable dose, orally Q2D with 28 days each cycle

SUMMARY:
This is a Phase 1, first-in-human, open-label study of JAB-8263 to determine the maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D) and assess the DLT. 30 subjects with advanced solid tumor will be enrolled.

DETAILED DESCRIPTION:
JAB-8263 is a small-molecule inhibitor of the highly conserved bromodomain pockets of the bromodomain and extraterminal (BET) proteins.

The objectives of this study are:

To determine the maximum-tolerated dose (MTD) and assess the dose-limiting toxicity (DLT) of JAB-8263 as a single agent to adult subjects with advanced solid tumors To assess the safety and tolerability of JAB-8263 To characterize the pharmacokinetic (PK) parameters and pharmacodynamics (PDc) To evaluate preliminary antitumor activity of JAB-8263

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria in order to be included in the research study:

1. Subject must be ≥18 years-of-age at the time of signature of the informed consent form (ICF).
2. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
3. Subjects with histologically or cytologically confirmed advanced solid tumors which have progressed despite standard therapy(ies), or are intolerant to standard therapy(ies), or have a tumor for which no standard therapy(ies) exists.
4. Subjects with life expectancy ≥3 months.
5. Patients must have at least one measurable lesion as defined by RECIST v1.1.
6. Patients who have sufficient baseline organ function.

Exclusion Criteria:

1. History (≤3 years) of cancer that is histologically distinct from the cancer under study.
2. Known serious allergy to investigational drug or excipients
3. Active brain or spinal metastases
4. History of pericarditis or Grade ≥2 pericardial effusion
5. History of interstitial lung disease.
6. History of Grade ≥2 active infections within 2 weeks
7. Known human immunodeficiency virus (HIV) infection
8. Seropositive for hepatitis B virus (HBV)
9. Seropositive for hepatitis C virus (HCV), or HCV-RNA viral levels are not detectable.
10. Any severe and/or uncontrolled medical conditions
11. History of myocardial infarction, unstable angina pectoris, coronary artery bypass graft, or cerebrovascular accident
12. Impaired cardiac function or clinically significant cardiac diseases
13. QTcF >470 msec at screening
14. History of medically significant thromboembolic events or bleeding diathesis
15. Unresolved Grade >1 toxicity
16. History of malignant biliary obstruction
17. Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | Approximately 2.5 years
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle with JAB-8263
Find Recommended Phase 2 Dose (RP2D) of JAB-8263 | Approximately 2.5 years
  Measurements of MTD (i.e. the highest dose of JAB-8263 associated with the occurrence of Dose Limiting Toxicities (DLTs) in <33% of patients) or the RP2D (i.e. the highest tested dose that is declared safe and tolerable by the Investigators and Sponsor)

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 2.5 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments
Area under the curve | Approximately 2.5 years
  Area under the plasma concentration time curve of JAB-8263
Cmax | Approximately 2.5 years
  Highest observed plasma concentration of JAB-8263
Tmax | Approximately 2.5 years
  Time of highest observed plasma concentration of JAB-8263
T1/2 | Approximately 2.5 years
  Half life of JAB-8263
Objective response rate ( ORR ) | Approximately 2.5 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Duration of response ( DOR ) | Approximately 2.5 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobio Pharmaceuticals, Study Director — Jacobio Pharmaceuticals
Locations (3):
- United States (3):
  - SCRI HeatlthONE, Denver, Colorado
  - Florida Cancer Center, Lake Mary, Lake City, Florida
  - Tennessee Oncology Nashville, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No